CLINICAL TRIAL: NCT04547270
Title: High Definition Ultrasound Imaging of the Intermuscular Bridges at the Interscalene Groove: A Prospective Observational Volunteer Study
Brief Title: High Definition Ultrasound Imaging of the Intermuscular Bridges at the Interscalene Groove
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof Manoj K Karmakar, Professor, Chinese University of Hong Kong
Other Study IDs: Intersca Vol Scan 2020.356
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Healthy
Keywords: interscalene groove; intermuscular bridges
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrasound scan — Volunteers will have an ultrasound scanning of both sides of their neck lying in supine position. Sequentially the scanning will start from the base of the neck (supraclavicular fossa) to the upper part of the interscalene groove and then in the reverse direction to the supraclavicular fossa. Images will be recorded as video loops.

SUMMARY:
This study aims to define the intermuscular bridges between the scalene muscles at the interscalene groove (around neck area) using high definition US imaging in a cohort of volunteers.

DETAILED DESCRIPTION:
The Interscalene brachial plexus block (ISBPB), with recent techniques like phrenic nerve sparing interscalene approach, has better safety profile than before and because of this, it is often the technique of choice for anaesthesia and/or analgesia during shoulder and proximal arm surgery. Anatomical variations at the interscalene groove are not uncommon and few have been described in the literature. Understanding the anatomy of the brachial plexus and its sheath at the interscalene groove is vital for the success of the block and to reduce the risk of complications during ultrasound (US) guided ISBPB. Recently, with the use of high definition ultrasound, using high frequency linear transducer, the principal investigator have identified intermuscular bridges appearing between the ventral rami of the brachial plexus at the interscalene groove. These intermuscular bridges may affect the spread of local anesthetic dispersion within the brachial plexus sheath thereby affecting the block dynamics of ISBPB. Therefore, this prospective observational study aim to define the intermuscular bridges at the interscalene groove using high definition ultrasound imaging in a group of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* volunteers consented for the scanning

Exclusion Criteria:

* prior surgery on either side of the neck
* presence of obvious deformity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult volunteers among staff, residents and their friends
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of the interscalene muscular ridges | through study completion, an average of 20 minutes.
  Volunteers will have ultrasound (USG) scanning of both sides of their necks that last for 20 minutes. Images will be recorded as video loops of 7 seconds each that include supraclavicular fossa, C5-7 transverse processes, superior, middle and inferior trunk. After completion of all scannings, newly coded video loops not in a predetermined order or sequence, will be assessed by 3 senior anaesthesiologists and the visualization of the intermuscular bridges at the interscalene groove will be noted. The quality of ultrasound visibility (ultrasound visibility score, UVS) of each structure will be assessed using a 4-point Likert scale (0, not visible; 1, hardly visible; 2, well visible; 3, very well visible). Total UVS (maximum score possible=15) will be calculated by averaging the scores from the three outcome assessors. The percentage of agreement among 3 outcome assessors will be determined by using data on positive identification of the interscalene muscular ridges.

CONTACTS AND LOCATIONS:
Overall Officials: Manoj K Karmakar, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Kowloon, Hong Kong